CLINICAL TRIAL: NCT01691352
Title: Prospective, Randomized Controlled Trial of Wound Management After Ostomy Closure
Brief Title: Wick vs. No Wick: Does Method of Closure Affect Rate of Wound Infection?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of sufficient population for recruitment
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stoma Closure_Wound Infection
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Wound Infection
Keywords: Wound infection; Ostomy reversal
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wick (Active Comparator): Patients with wick placed in their wound at the time of ostomy reversal
  Interventions: Procedure: Wick dressing
- No wick (Sham Comparator): patients with non-wicked dressing placed on their wound
  Interventions: Procedure: No Wick

INTERVENTIONS:
Procedure: Wick dressing — Once the fascia of the ostomy site is closed, the subcutaneous space will be irrigated with normal saline. The skin will then be reapproximated using an absorbable suture, spaced every 1 cm across the wound (i.e. for a 2cm wound, a single suture will be placed in the middle). A moist, saline/betadine soaked gauze will then be gently packed into the wound spaces, on either side of the sutures. The gauze will be packed into the wound to the depth of ½ a cm, or ½ of the wound depth, whichever is greater. A single dry piece of gauze will then be secured over the top of the wound. Dressings and packing will be removed by the surgical team on post-operative day 2
  Arms: Wick
Procedure: No Wick — Once the fascia of the ostomy site is closed, the subcutaneous space will be irrigated with normal saline. The skin will then be reapproximated using an absorbable suture, spaced every 1 cm across the wound (i.e. for a 2 cm wound, a single suture will be placed in the middle). A single piece of dry gauze will then be secured over the top of the wound. Dressings will be removed by the surgical team on post-operative day 2
  Arms: No wick

SUMMARY:
Countless children undergo surgery annually for management of what clinicians consider to be a "dirty wound". One frequently encountered example is the ostomy reversal. During this planned operation, the previously diverted small bowel or colon is reconnected with the distal intestine, restoring continuity. However, this procedure leaves an open wound on the anterior abdominal wall, creating a conundrum for the surgeon and raises the question: how should the wound be managed? In the investigators practice at CHOA, surgeons utilize both a wick and a non-wicked wound dressing. In this prospective randomized trial, we wish to evaluate these two dressings in children receiving an ostomy closure. The investigators hypothesis is that the incidence of wound infection after ostomy reversal is the same regardless of if a wick is placed or not.

DETAILED DESCRIPTION:
Countless children undergo surgery annually for management of what clinicians consider to be a "dirty wound". These include any case where the patient has a known intraabdominal infection or enteric contents are likely to have contaminated the surgical field. One frequently encountered example is the ostomy reversal. During this planned operation, the previously diverted small bowel or colon is reconnected with the distal intestine, restoring continuity. However, this procedure leaves an open wound on the anterior abdominal wall, creating a conundrum for the surgeon and raises the question: how should the wound be managed?

Historically, surgeons would close the ostomy site in a primary fashion using a running subcuticular suture. While there is no "national standard" for wound closure of ostomies, concern over the likelihood of local wound infection has led most modern day practitioners to leave the wound open to drain in some fashion. Still the techniques used varies from the use of simple interrupted sutures along the wound incision to the use of a betadine soaked gauze "wick" in the wound. Other surgeons have attempted to close ostomy sites in a delayed fashion, 48-72 hours after the primary operation.

Limited research has been prospectively performed to evaluate and compare the merit of these techniques. In children, there has been no recent data directly addressing this question.

In our practice at CHOA, surgeons utilize both a wick and a non-wicked wound dressing. Our current wound infection rate is approximately 10%, defined as spreading redness, draining pus, fever, increased wound tenderness in the perioperative period. Unfortunately, the type of dressing placed at the end of an operation is rarely, if ever documented in an operative note, therefore a retrospective review to assess outcomes is not feasible. While there is no exact statistics for how many ostomies were closed using a wick versus an non-wicked dressing, in a survey of our 7 physicians, approximately 50% of the attending report that they place a wick on all of their patients and the remaining attendings do not use a wick with the rare exception of a particularly "dirty wound" (i.e. significant spillage of stool into the wound or grossly necrotic/infected tissue) or a particularly deep wound. Clinicians who elect to use a wick have adopted that practice based on person opinion that it allows the wounds to drain better, thus preventing infection. Those who do not place a wick state that they feel it is an unnecessary step in the dressing and that interrupted sutures alone are sufficient to allow the wound to drain.

After a lengthy discussion with all of the surgeons at Egleston and 4 of the surgeons at Scottish Rite, as a department, we have decided to evaluate the type of dressing used for ostomy closure in order to see if there is in fact any benefit to leaving a wick in the ostomy wound. All of the surgeons have agreed to participate in this study without undo bias.

In this prospective randomized trial, we wish to evaluate these two dressings in children receiving an ostomy closure. Our hypothesis is that the incidence of wound infection after ostomy reversal is the same regardless of if a wick is placed or not.

ELIGIBILITY:
Inclusion Criteria:

All patients at Children's Healthcare of Atlanta (Egleston or Scotish Rite campus) who are scheduled to undergo an ostomy reversal will be approached for participation in this study. As there truly is no known "better" dressing for this type of wound, all patients, including those with co-morbidities such as immunosuppression will be eligible for inclusion in this study. Only those whose families consent to be included in the study will be included or randomized to the study.

Exclusion Criteria:

Patients who do not give consent to participate will be excluded from this study. Additionally, if at the time of the operation, the surgeon feels that it is not in the patient's best interest to be randomized and included in the study, he/she may decide to exclude the patient.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Wound infection | 14 days
  We will be evaluating wound infection rate, as determined by spreading redness, draining pus, fever, increased wound tenderness in the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Clifton, MD, Principal Investigator — Faculty Surgeon
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States